CLINICAL TRIAL: NCT06505512
Title: A Study on the Significance of Joint Evaluation of Gastrointestinal Ultrasound Results and Renal Artery Resistance Index for Assessing the Intestinal-renal Syndrome in Sepsis Patients
Brief Title: A Study of Enterorenal Syndrome Assessed by Gastrointestinal Ultrasound Combined with Renal Artery Resistance Index
Status: Recruiting | Type: Observational
Sponsor: Zhangzhou Municipal Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: zqj123456
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-07

CONDITIONS: Sepsis; Urinary Tract Infections
MeSH Terms: conditions — Sepsis; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Survival group: Patients who get better after treatment and eventually survive.
  Interventions: Diagnostic Test: No intervention
- Death group: Patients who die within 28 days of hospitalization.
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
In this study, the patients with sepsis caused by abdominal infection were divided into survival group and death group by ultrasound examination of gastrointestinal function, superior mesenteric artery blood flow, and renal artery resistance index. The cross-sectional area of gastric antrum, average time flow rate of superior mesenteric artery, colon diameter, colon peristalsis frequency, and renal artery resistance index of the two groups were compared to determine the progression of entero-renal syndrome as soon as possible. To provide reliable objective basis for clinical decision-making, in order to improve the success rate of rescue.

DETAILED DESCRIPTION:
Adult patients admitted to EICU of our hospital who met the diagnostic criteria for sepsis were included in the study. Patients with intra-abdominal sepsis were divided into survival group and death group for case control. Exclusion criteria: open chest and abdomen injury, advanced tumor, uremia, pregnancy. The primary endpoint was survival. Extraction time: ICU (0h), ICU (6h, that is, after fluid resuscitation), ICU (24h), ICU (48h, 08:00 a.m.), ICU (72h, 08:00 a.m.), ICU (120h, 08:00 a.m.); Monitoring indicators: antral cross-section area, colon diameter, colon peristalsis frequency, renal artery resistance index, CVP, ScvO2, IL6, blood lactic acid, blood creatinine, fluid intake, bladder pressure. The primary endpoint of the study was survival rate, and statistical analysis was performed to evaluate the progression of enterorenal syndrome, provide reliable objective basis for subsequent clinical decision-making, and improve the success rate of rescue.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with intra-abdominal infections
* Patients with sepsis or septic shock

Exclusion Criteria:

* Patients with open chest or abdominal injury
* Patients with advanced tumor
* Patients with uremia
* Pregnant women

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this study, patients who had been admitted into the ICU of our hospital due to sepsis/spetic shock induced by intra-abdominal infections and who had stayed for more than 72 hours.The patients with sepsis caused by abdominal infection were divided into survival group and death group by ultrasound examination of gastrointestinal function, superior mesenteric artery blood flow, and renal artery resistance index. The cross-sectional area of gastric antrum, average time flow rate of superior mesenteric artery, colon diameter, colon peristalsis frequency, and renal artery resistance index of the two groups were compared to determine the progression of entero-renal syndrome as soon as possible.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
superior mesenteric artery resistance index | upon admission into the ICU, and, 24 and 72 hours afterwards
  With the patient in a supine position, ran the probe along the longitudinal section of the abdominal aorta to reveal the long axis of the superior mesenteric artery, and placed the probe 1.0 to 2.0 cm distal of where the superior mesenteric artery starts. The pulsed wave Doppler was used to show the spectrum of blood flow velocity, where the included angle between the bloodstream and the sound beam ranged from 25° to 45°. The waveform was recorded for three cardiac cycles, and the mean value calculated(Figure 1). The normal value of SMARI was between 0.69~0.91
renal artery resistance index | upon admission into the ICU, and, 24 and 72 hours afterwards
  With the patient in a supine position, ran the probe along the longitudinal section of the abdominal aorta to reveal the long axis of the superior mesenteric artery, and placed the probe 1.0 to 2.0 cm distal of where the superior mesenteric artery starts. The pulsed wave Doppler was used to show the spectrum of blood flow velocity, where the included angle between the bloodstream and the sound beam ranged from 25° to 45°. The waveform was recorded for three cardiac cycles, and the mean value calculated(Figure 1). The normal value of SMARI was between 0.69~0.91

CONTACTS AND LOCATIONS:
Overall Officials: Hui Jiang, Dr., Principal Investigator — the Ethnics Committee of Zhangzhou Municipal Hospital of Fujian Province
Locations (1):
- Qingjiang Zheng, Zhangzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No